CLINICAL TRIAL: NCT00081224
Title: A Phase II Trial Of Celecoxib (Celebrex) And Capecitabine (Xeloda) Combined With Pelvic Irradiation As Neoadjuvant Treatment Of Stage II or III Adenocarcinoma Of The Rectum
Brief Title: Neoadjuvant Celecoxib and Capecitabine Combined With Pelvic Irradiation in Treating Patients With Stage II or Stage III Adenocarcinoma (Cancer) of the Rectum
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0346; NCI-2012-02582 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000360666 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the rectum; stage II rectal cancer; stage III rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Celecoxib; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- celecoxib + capecitabine + radiation + surgery (Experimental): Neoadjuvant chemoradiotherapy: Patients receive oral celecoxib twice daily on days 1-7 and oral capecitabine twice daily on days 1-5. Patients undergo pelvic radiotherapy once daily on days 1-5. Courses repeat weekly for 5.5 weeks.
  Surgery: Patients undergo surgery 4-6 weeks after completion of neoadjuvant chemoradiotherapy.
  Adjuvant chemotherapy: Patients with a curative resection receive oral capecitabine twice daily on days 1-14. Treatment repeats every 21 days for up to 4 courses.
  Treatment continues in the absence of disease progression or unacceptable toxicity.
  Patients are followed every 3 months for 1 year and then every 6 months for 4 years.
  Interventions: Drug: capecitabine; Drug: celecoxib; Radiation: radiation therapy; Procedure: surgery

INTERVENTIONS:
Drug: capecitabine
Drug: celecoxib
Radiation: radiation therapy
Procedure: surgery

SUMMARY:
RATIONALE: Celecoxib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Drugs used in chemotherapy, such as capecitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Celecoxib may also make tumor cells more sensitive to chemotherapy and radiation therapy. Giving celecoxib with capecitabine and radiation therapy before surgery may shrink the tumor so that it can be removed.

PURPOSE: This phase II trial is studying how well giving neoadjuvant celecoxib together with capecitabine and pelvic irradiation works in treating patients with stage II or stage III adenocarcinoma (cancer) of the rectum.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the pathological complete response rate in patients with stage II or III adenocarcinoma of the rectum treated with neoadjuvant celecoxib and capecitabine in combination with pelvic irradiation.

Secondary

* Determine the safety and tolerability of this regimen in these patients.
* Determine the rectal function of patients treated with this regimen.
* Determine the time to recurrence or progression and survival time of patients treated with this regimen.
* Correlate cellular and molecular markers in pretreatment tumor samples with response in patients treated with this regimen.

OUTLINE: This is a multicenter study.

* Neoadjuvant chemoradiotherapy: Patients receive oral celecoxib twice daily on days 1-7 and oral capecitabine twice daily on days 1-5. Patients undergo pelvic radiotherapy once daily on days 1-5. Courses repeat weekly for 5.5 weeks.
* Surgery: Patients undergo surgery 4-6 weeks after completion of neoadjuvant chemoradiotherapy.
* Adjuvant chemotherapy: Patients with a curative resection receive oral capecitabine twice daily on days 1-14. Treatment repeats every 21 days for up to 4 courses.

Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year and then every 6 months for 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed rectal adenocarcinoma

  * Clinical stage T3, N0, M0 OR any T, N1-3, M0 disease
* Treatment with neoadjuvant chemotherapy and pelvic radiotherapy is indicated

  * All disease must be encompassable within standard pelvic radiotherapy fields
* Distal border of the tumor must be at or below* the peritoneal reflection, defined as within 12 cm of the anal verge by endoscopy NOTE: *If a portion of the tumor is below the peritoneal reflection at the time of surgery, patients are eligible regardless of the distance of the tumor determined at endoscopy
* Tumor must be determined to be clinically resectable

  * Tumor may not be clinically fixed
  * Negative margins by routine examination of an unanesthetized patient
* Transmural penetration of tumor through the muscularis propria by CT scan, endorectal ultrasound, or MRI
* No distant metastatic disease

  * No evidence of tumor outside the pelvis, including any of the following:

    * Metastatic inguinal lymphadenopathy
    * Peritoneal seeding
    * Liver metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* At least 6 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ upper limit of normal (ULN)
* AST ≤ 3 times ULN
* Alkaline phosphatase ≤ 4 times ULN if AST < ULN

Renal

* Creatinine clearance ≥ 30 mL/min
* No renal impairment

Cardiovascular

* No congestive heart failure
* No symptomatic coronary artery disease
* No uncontrolled cardiac arrhythmias
* No myocardial infarction
* No history of transient ischemic attacks or stroke
* No other clinically significant cardiac disease

Gastrointestinal

* No bleeding peptic ulcer disease within the past 12 months
* No lack of physical integrity of the upper gastrointestinal tract
* No malabsorption syndrome
* No active inflammatory bowel disease
* Must be able to swallow study drugs

Other

* No dihydropyrimidine dehydrogenase deficiency
* No history of uncontrolled seizures
* No CNS disorders
* No clinically significant psychiatric illness that would preclude study compliance or giving informed consent
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No known sensitivity to NSAIDs, sulfonamides, or aspirin
* No other serious medical illness that would preclude study treatment
* No other conditions that would preclude study participation
* Must be able to tolerate major surgery that may include abdominal-perineal resection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 30 days after study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No prior systemic anticancer chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* No prior radiotherapy to the pelvis

Surgery

* See Disease Characteristics
* More than 3 weeks since prior major surgery and recovered

Other

* At least 7 days since prior nonsteroidal anti-inflammatory drugs (NSAIDs), including aspirin
* No other concurrent investigational drugs
* No other concurrent anticancer treatment
* No concurrent NSAIDs
* No concurrent primary prophylactic therapy for hand-foot syndrome
* No concurrent loperamide prophylaxis for diarrhea
* No concurrent sorivudine or brivudine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2004-12; Primary Completion 2006-02 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Proportion of successes | Up to 5 years

SECONDARY OUTCOMES:
Survival time | Up to 5 years
Time-to event analyses | Up to 5 years
Time to disease progression/recurrence | Up to 5 years
Time to recurrence | Up to 5 years
Time to first progression | Up to 5 years
Survival | Up to 5 years
Bowel function as measured by the Patient Bowel Function (Uniscale) Questionnaire, the FACT Diarrhea Subscale and the Mayo Bowel Function Questionnaire | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Frank Sinicrope, MD, Study Chair — Mayo Clinic